CLINICAL TRIAL: NCT02416193
Title: Can Vitamin D3 Improve Cognitive Function in Individuals With Type 2 Diabetes? (THINK-D)
Acronym: THINK-D
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study was halted prematurely due to slow recruitment and expiration of funding
Sponsor: Loyola University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Mary A Byrn, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206988; 206988031815 (Other: Loyola University Chicago)
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Diabetes; Executive Dysfunction
Keywords: Diabetes; Cognition; Functioning
MeSH Terms: conditions — Diabetes Mellitus | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose (Experimental): 50,000 IU cholecalciferol once weekly for three months
  Interventions: Drug: Cholecalciferol
- Low Dose (Active Comparator): 5,000 IU cholecalciferol once weekly for three months
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Participants will take randomly assigned high dose cholecalciferol once weekly for three months
  Other Names: Vitamin D3
  Arms: High Dose
Drug: Cholecalciferol — Participants will take randomly assigned active comparator cholecalciferol once weekly for three months
  Other Names: Vitamin D3
  Arms: Low Dose

SUMMARY:
Diabetes increases the risk of cognitive dysfunction. The incidence of dementia is 1.5 to 2.5 times higher in persons with diabetes than the general population. There is evidence that cognitive decline significantly impacts the ability to self-manage diabetes. Strategies to prevent cognitive decline in persons with diabetes has not been well studied. A recent study reported that in persons who had vitamin D deficiency, the risk for all-cause dementia and Alzheimer's was doubled. Vitamin D receptors are located in the brain and deficiency of vitamin D has been reported to negatively affect the development of brain. Therefore, providing vitamin D supplementation to improve cognitive function is worthy of study. The investigators propose a small, randomized controlled trial to determine the effects of vitamin D3 supplementation in persons with type 2 diabetes who have symptoms of cognitive impairment. Persons will be randomized to receive either weekly vitamin D3 supplementation (50,000 IUs) or a matching comparator (5000 IUs) for a period of three months. The study aims are to determine (1) the effect of vitamin D3 supplementation on cognitive function and (2) the effect of vitamin D3 supplementation on diabetes self-management. A sample of persons with type 2 diabetes (n=62), who have a subjective complaint of a cognitive dysfunction or scoring at least one standard deviation below normal on a cognitive functioning screening test, have vitamin D levels less 30 ng/ml, are not depressed (as this impacts cognitive function), and do not have severe diabetes complication will be recruited. Participants will be phone screened and complete two baseline visits prior to randomization. They will then have phone call and follow-up visits to assess (1) cognitive function using standardized tests to assess for executive function (2) serum measurements (HBA1c, fasting glucose, vitamin D levels, and cardiometabolic profile) and (3) surveys to assess cognitive function as well as self-management behaviors.

DETAILED DESCRIPTION:
Study Aims Diabetes increases the risk of cognitive dysfunction. The incidence of dementia is 1.5 to 2.5 times higher in persons with diabetes than the general population (1). There is evidence that cognitive decline significantly impacts the ability to self-manage diabetes (2). Strategies to prevent cognitive decline in persons with diabetes has not been well studied. A recent study reported that in persons who had vitamin D deficiency, the risk for all-cause dementia and Alzheimer's was doubled (3). Vitamin D receptors are located in the brain, and deficiency of vitamin D has been reported to negatively affect the development of brain and impact both growth factor signaling and neural activity (4, 5). Therefore, providing vitamin D supplementation to improve cognitive function in persons with diabetes who are at great risk for this comorbid condition is important. The investigators propose a small, randomized controlled trial to determine the effects of vitamin D3 supplementation in persons with type 2 diabetes who have symptoms of cognitive impairment. Persons will be randomized to receive either weekly vitamin D3 supplementation (50,000 IUs) or a matching comparator (5000 IUs) for a period of three months.

Primary Aim: To determine the effect of vitamin D3 supplementation on cognitive function for persons with type 2 diabetes.

Primary Hypothesis: Persons receiving weekly vitamin D3 supplementation (50,000 IUs) will have improved cognitive function compared to those receiving the comparator (5000 IUs) at three months.

Secondary Aim: To determine the effect of vitamin D3 supplementation on diabetes self-management.

Secondary Hypothesis: Persons receiving weekly vitamin D3 supplementation (50,000 IUs) will have improved self-management compared to those receiving the comparator (5000 IUs) at three months.

The importance of this study is several fold. Vitamin D supplementation is a low cost intervention (6), it has minimal side effects (7), and it could have high impact for persons with type 2 diabetes who suffer from cognitive impairment which can significantly affect their diabetes self-management.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 to 75 years
* Have type 2 diabetes
* Having a subjective complaint of a cognitive dysfunction or scoring at least one standard deviation below normal on a cognitive functioning screening test
* Vitamin D level as measured by 25-hydroxyvitamin D (25-OH D) < 32 ng/mL
* Under the care of a healthcare provider
* Systolic blood pressure ≤160 and diastolic blood pressure ≤100

Exclusion Criteria:

* Persons with malabsorption problems (e.g., crohn's disease)
* Hypercalcemia
* Supplementation other than a daily multivitamin
* Severe complications of diabetes (i.e., amputation, blindness, and dialysis)
* Concomitant use of steroids
* GFR < 60
* Creatinine > 1.2
* Significant depressive symptoms
* Having a history of bipolar depression, psychotic disorders, loss of consciousness greater than 5 minutes, or a current alcohol or substance use disorder
* Other serious medical conditions deemed significant by the PI or medical monitor
* Concomitant use of cholinesterase inhibitors
* Concomitant use of anxiolytics, kava kava, St. John's Wort, or Ginkgo Biloba
* Pregnancy
* HbA1c >13%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Byrn, Ph.D., R.N., Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers

REFERENCES:
- [Background] Lee JH, Choi Y, Jun C, Hong YS, Cho HB, Kim JE, Lyoo IK. Neurocognitive changes and their neural correlates in patients with type 2 diabetes mellitus. Endocrinol Metab (Seoul). 2014 Jun;29(2):112-21. doi: 10.3803/EnM.2014.29.2.112. PMID 25031883
- [Background] Smith MA, Else JE, Paul L, Foster JK, Walker M, Wesnes KA, Riby LM. Functional Living in Older Adults With Type 2 Diabetes: Executive Functioning, Dual Task Performance, and the Impact on Postural Stability and Motor Control. J Aging Health. 2014 Aug;26(5):841-859. doi: 10.1177/0898264314534896. Epub 2014 Jun 4. PMID 24898849
- [Background] Littlejohns TJ, Henley WE, Lang IA, Annweiler C, Beauchet O, Chaves PH, Fried L, Kestenbaum BR, Kuller LH, Langa KM, Lopez OL, Kos K, Soni M, Llewellyn DJ. Vitamin D and the risk of dementia and Alzheimer disease. Neurology. 2014 Sep 2;83(10):920-8. doi: 10.1212/WNL.0000000000000755. Epub 2014 Aug 6. PMID 25098535
- [Background] McCann JC, Ames BN. Is there convincing biological or behavioral evidence linking vitamin D deficiency to brain dysfunction? FASEB J. 2008 Apr;22(4):982-1001. doi: 10.1096/fj.07-9326rev. Epub 2007 Dec 4. PMID 18056830
- [Background] Schlogl M, Holick MF. Vitamin D and neurocognitive function. Clin Interv Aging. 2014 Apr 2;9:559-68. doi: 10.2147/CIA.S51785. eCollection 2014. PMID 24729696
- [Background] Holick MF. High prevalence of vitamin D inadequacy and implications for health. Mayo Clin Proc. 2006 Mar;81(3):353-73. doi: 10.4065/81.3.353. PMID 16529140
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Tuligenga RH, Dugravot A, Tabak AG, Elbaz A, Brunner EJ, Kivimaki M, Singh-Manoux A. Midlife type 2 diabetes and poor glycaemic control as risk factors for cognitive decline in early old age: a post-hoc analysis of the Whitehall II cohort study. Lancet Diabetes Endocrinol. 2014 Mar;2(3):228-35. doi: 10.1016/S2213-8587(13)70192-X. Epub 2013 Dec 19. PMID 24622753
- [Background] Wennberg AMV, Gottesman RF, Kaufmann CN, Albert MS, Chen-Edinboro LP, Rebok GW, Kasper JD, Spira AP. Diabetes and cognitive outcomes in a nationally representative sample: the National Health and Aging Trends Study. Int Psychogeriatr. 2014 Oct;26(10):1729-1735. doi: 10.1017/S1041610214001380. Epub 2014 Jul 30. PMID 25075535
- [Background] Munshi MN, Hayes M, Iwata I, Lee Y, Weinger K. Which aspects of executive dysfunction influence ability to manage diabetes in older adults? Diabet Med. 2012 Sep;29(9):1171-7. doi: 10.1111/j.1464-5491.2012.03606.x. PMID 22340082
- [Background] Grober E, Hall CB, Hahn SR, Lipton RB. Memory Impairment and Executive Dysfunction are Associated with Inadequately Controlled Diabetes in Older Adults. J Prim Care Community Health. 2011 Oct 1;2(4):229-33. doi: 10.1177/2150131911409945. Epub 2011 Jun 1. PMID 23804840
- [Background] Retracted: Executive dysfunction in elderly diabetic patients. Geriatr Gerontol Int. 2015 Aug;15(8):1106. doi: 10.1111/ggi.12288. Epub 2014 Apr 21. No abstract available. PMID 24750335
- [Background] Winkler A, Dlugaj M, Weimar C, Jockel KH, Erbel R, Dragano N, Moebus S. Association of diabetes mellitus and mild cognitive impairment in middle-aged men and women. J Alzheimers Dis. 2014;42(4):1269-77. doi: 10.3233/JAD-140696. PMID 25024326
- [Background] Geijselaers SLC, Sep SJS, Stehouwer CDA, Biessels GJ. Glucose regulation, cognition, and brain MRI in type 2 diabetes: a systematic review. Lancet Diabetes Endocrinol. 2015 Jan;3(1):75-89. doi: 10.1016/S2213-8587(14)70148-2. Epub 2014 Aug 24. PMID 25163604
- [Background] Annweiler C, Montero-Odasso M, Llewellyn DJ, Richard-Devantoy S, Duque G, Beauchet O. Meta-analysis of memory and executive dysfunctions in relation to vitamin D. J Alzheimers Dis. 2013;37(1):147-71. doi: 10.3233/JAD-130452. PMID 23948884
- [Background] Penckofer S, Kouba J, Wallis DE, Emanuele MA. Vitamin D and diabetes: let the sunshine in. Diabetes Educ. 2008 Nov-Dec;34(6):939-40, 942, 944 passim. doi: 10.1177/0145721708326764. PMID 19075078
- [Background] Gulseth HL, Gjelstad IM, Tierney AC, Lovegrove JA, Defoort C, Blaak EE, Lopez-Miranda J, Kiec-Wilk B, Riserus U, Roche HM, Drevon CA, Birkeland KI. Serum vitamin D concentration does not predict insulin action or secretion in European subjects with the metabolic syndrome. Diabetes Care. 2010 Apr;33(4):923-5. doi: 10.2337/dc09-1692. Epub 2010 Jan 12. PMID 20067973
- [Background] Davidson MB, Duran P, Lee ML, Friedman TC. High-dose vitamin D supplementation in people with prediabetes and hypovitaminosis D. Diabetes Care. 2013 Feb;36(2):260-6. doi: 10.2337/dc12-1204. Epub 2012 Oct 1. PMID 23033239
- [Background] Penckofer S, Kouba J, Byrn M, Estwing Ferrans C. Vitamin D and depression: where is all the sunshine? Issues Ment Health Nurs. 2010 Jun;31(6):385-93. doi: 10.3109/01612840903437657. PMID 20450340
- [Background] Drechsler C, Schmiedeke B, Niemann M, Schmiedeke D, Kramer J, Turkin I, Blouin K, Emmert A, Pilz S, Obermayer-Pietsch B, Weidemann F, Breunig F, Wanner C. Potential role of vitamin D deficiency on Fabry cardiomyopathy. J Inherit Metab Dis. 2014 Mar;37(2):289-95. doi: 10.1007/s10545-013-9653-8. Epub 2013 Oct 19. PMID 24141790
- [Background] Alves MR, Yamamoto T, Arias-Carrion O, Rocha NB, Nardi AE, Machado S, Silva AC. Executive function impairments in patients with depression. CNS Neurol Disord Drug Targets. 2014;13(6):1026-40. doi: 10.2174/1871527313666140612102321. PMID 24923347
- [Background] Zahodne LB, Nowinski CJ, Gershon RC, Manly JJ. Depressive symptoms are more strongly related to executive functioning and episodic memory among African American compared with non-Hispanic White older adults. Arch Clin Neuropsychol. 2014 Nov;29(7):663-9. doi: 10.1093/arclin/acu045. Epub 2014 Oct 3. PMID 25280795
- [Background] Jorde R, Sneve M, Figenschau Y, Svartberg J, Waterloo K. Effects of vitamin D supplementation on symptoms of depression in overweight and obese subjects: randomized double blind trial. J Intern Med. 2008 Dec;264(6):599-609. doi: 10.1111/j.1365-2796.2008.02008.x. Epub 2008 Sep 10. PMID 18793245
- [Background] Burton JM, Kimball S, Vieth R, Bar-Or A, Dosch HM, Cheung R, Gagne D, D'Souza C, Ursell M, O'Connor P. A phase I/II dose-escalation trial of vitamin D3 and calcium in multiple sclerosis. Neurology. 2010 Jun 8;74(23):1852-9. doi: 10.1212/WNL.0b013e3181e1cec2. Epub 2010 Apr 28. PMID 20427749
- [Background] Nazarian S, St Peter JV, Boston RC, Jones SA, Mariash CN. Vitamin D3 supplementation improves insulin sensitivity in subjects with impaired fasting glucose. Transl Res. 2011 Nov;158(5):276-81. doi: 10.1016/j.trsl.2011.05.002. Epub 2011 Jun 7. PMID 22005267
- [Background] Recker RR, Gallagher R, MacCosbe PE. Effect of dosing frequency on bisphosphonate medication adherence in a large longitudinal cohort of women. Mayo Clin Proc. 2005 Jul;80(7):856-61. doi: 10.4065/80.7.856. PMID 16007889
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Mitri J, Dawson-Hughes B, Hu FB, Pittas AG. Effects of vitamin D and calcium supplementation on pancreatic beta cell function, insulin sensitivity, and glycemia in adults at high risk of diabetes: the Calcium and Vitamin D for Diabetes Mellitus (CaDDM) randomized controlled trial. Am J Clin Nutr. 2011 Aug;94(2):486-94. doi: 10.3945/ajcn.111.011684. Epub 2011 Jun 29. PMID 21715514
- [Background] Koutkia P, Lu Z, Chen TC, Holick MF. Treatment of vitamin D deficiency due to Crohn's disease with tanning bed ultraviolet B radiation. Gastroenterology. 2001 Dec;121(6):1485-8. doi: 10.1053/gast.2001.29686. PMID 11729127
- [Background] Lips P. Which circulating level of 25-hydroxyvitamin D is appropriate? J Steroid Biochem Mol Biol. 2004 May;89-90(1-5):611-4. doi: 10.1016/j.jsbmb.2004.03.040. PMID 15225848
- [Background] Etgen T, Sander D, Bickel H, Sander K, Forstl H. Vitamin D deficiency, cognitive impairment and dementia: a systematic review and meta-analysis. Dement Geriatr Cogn Disord. 2012;33(5):297-305. doi: 10.1159/000339702. Epub 2012 Jul 2. PMID 22759681
- [Background] Wallis DE, Penckofer S, Sizemore GW. The "sunshine deficit" and cardiovascular disease. Circulation. 2008 Sep 30;118(14):1476-85. doi: 10.1161/CIRCULATIONAHA.107.713339. No abstract available. PMID 18824654
- [Background] Glanz K, Yaroch AL, Dancel M, Saraiya M, Crane LA, Buller DB, Manne S, O'Riordan DL, Heckman CJ, Hay J, Robinson JK. Measures of sun exposure and sun protection practices for behavioral and epidemiologic research. Arch Dermatol. 2008 Feb;144(2):217-22. doi: 10.1001/archdermatol.2007.46. PMID 18283179
- [Background] Cummings SR, Block G, McHenry K, Baron RB. Evaluation of two food frequency methods of measuring dietary calcium intake. Am J Epidemiol. 1987 Nov;126(5):796-802. doi: 10.1093/oxfordjournals.aje.a114716. PMID 3661527
- [Background] Welch G, Weinger K, Anderson B, Polonsky WH. Responsiveness of the Problem Areas In Diabetes (PAID) questionnaire. Diabet Med. 2003 Jan;20(1):69-72. doi: 10.1046/j.1464-5491.2003.00832.x. PMID 12519323
- [Background] Ruff RM, Light RH, Parker SB, Levin HS. Benton Controlled Oral Word Association Test: reliability and updated norms. Arch Clin Neuropsychol. 1996;11(4):329-38. PMID 14588937
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gameroff MJ, Wickramaratne P, Weissman MM. Testing the Short and Screener versions of the Social Adjustment Scale-Self-report (SAS-SR). Int J Methods Psychiatr Res. 2012 Mar;21(1):52-65. doi: 10.1002/mpr.358. Epub 2011 Dec 5. PMID 22139969
- [Background] Endicott J, Nee J. Endicott Work Productivity Scale (EWPS): a new measure to assess treatment effects. Psychopharmacol Bull. 1997;33(1):13-6. PMID 9133746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place at Loyola University Medical Center (Maywood, IL) between September 2015 and June 2018
Pre-assignment Details: Fifty-six participants consented to participate in the study. Among these individuals, 26 (46.43%) were not randomized and were excluded from continuing their participation in the study because the medical monitor determined they did not meet study inclusion criteria.
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all individuals who consented to participate and took at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.62 (10.14) | 55.80 (9.68) | 55.71 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 9 | 17
  White | 5 | 4 | 9
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Years of education [Median (Inter-Quartile Range); unit: years] | 14 [12 to 15] | 14 [13 to 16] | 14 [13 to 15]
Total vitamin D level [Median (Inter-Quartile Range); unit: Nanograms per milliliter (ng/mL)] | 21 [15 to 25] | 25 [19 to 28] | 24 [17 to 27]
Serum vitamin D3 level [Median (Inter-Quartile Range); unit: Nanograms per milliliter (ng/mL)] | 21 [13 to 25] | 24 [18 to 28] | 22 [16 to 27]
Body mass index [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 40.44 (9.48) | 34.20 (5.05) | 37.32 (8.11)
Martial status [Count of Participants; unit: Participants]
  Currently married | 10 | 4 | 14
  Separated | 0 | 1 | 1
  Widowed | 2 | 0 | 2
  Divorced | 2 | 5 | 7
  Never married | 1 | 5 | 6
Season of first dose of the study drug [Count of Participants; unit: Participants]
  Fall | 5 | 5 | 10
  Winter | 3 | 6 | 9
  Spring | 5 | 1 | 6
  Summer | 2 | 3 | 5
Systolic blood pressure [Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)] | 134.73 (16.33) | 131.13 (16.95) | 132.93 (16.45)
Diastolic blood pressure [Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)] | 73.47 (10.99) | 72.93 (10.79) | 73.20 (10.70)
Heart rate [Mean (Standard Deviation); unit: Beats per minute (BPM)] | 73.27 (12.67) | 76.00 (12.86) | 74.63 (12.62)
HbA1c [Median (Inter-Quartile Range); unit: mmol/mol] | 7.10 [6.30 to 7.50] | 7.20 [6.20 to 7.80] | 7.15 [6.30 to 7.70]
Glucose [Median (Inter-Quartile Range); unit: Millimoles per liter (mmol/L)] | 120 [95 to 160] | 142 [116 to 214] | 134 [107 to 165]
Calcium [Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)] | 9.40 [9.30 to 9.60] | 9.60 [9.40 to 9.90] | 9.50 [9.30 to 9.70]
Creatinine [Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)] | 0.74 [0.66 to 0.90] | 0.83 [0.70 to 0.88] | 0.79 [0.69 to 0.88]
Activity level [Count of Participants; unit: Participants] — Baseline physical activity was assessed using the Godin Leisure-Time Exercise Questionnaire. The measure of physical activity ranges from 0 to infinity points. Scores less than 14 points on this assessment indicate insufficient physical activity while scores of 24 or higher indicate sufficient physical activity; other scores are categorized as being moderately active.
  Participants
    Insufficiently active | 5 | 6 | 11
    Moderately active | 3 | 3 | 6
    Sufficiently active | 7 | 6 | 13
WRAT-IV Reading Score [Median (Inter-Quartile Range); unit: units on a scale] — The Wide Range Achievement Test (WRAT-IV) reading subtest score is a 55-item assessment of letter and word decoding through letter identification and word recognition. Scores are standardized as z-scores using age-adjusted norms provided by Pearson Assessments (https://www.pearsonassessments.com/). A z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative z-scores indicate performance is lower than average, and positive z-scores indicate performance is higher than average. Positive z-scores indicate better performance.
  units on a scale | -1.00 [-1.20 to -0.33] | -0.93 [-1.20 to -0.20] | -0.97 [-1.20 to -0.33]
Patient Health Questionnaire-9 [Median (Inter-Quartile Range); unit: units on a scale] — The Patient Health Questionnaire-9 is an assessment of depression. Scores range from 1 to 27 points with higher scores indicating worse mood.
  units on a scale | 2 [1 to 4] | 4 [3 to 7] | 3 [2 to 5]
CES-D Score [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiologic Studies Depression (CES-D) assessment measures mood. Scores range from 0 to 60 points with higher scores indicating worse symptoms
  units on a scale | 7.13 (3.46) | 9.73 (4.80) | 8.43 (4.32)

OUTCOME MEASURES:

1. Primary Outcome: Letter-Number Sequencing
Description: The the Letter-Number Sequencing Test (from the Wechsler Adult Intelligence Scale-III assessment) is an assessment of working memory. Scores on the assessment are standardized as scaled scores with a mean of 10 and standard deviation of 3 (μ = 10, SD = 3) using age adjusted normative data provided by Pearson assessments (https://www.pearsonassessments.com/). A scaled score indicates the number of standard deviations away from the mean. A scaled score of 10 is equal to the mean. Scaled scores below 10 indicate performance is lower than average, and scaled scores higher than 10 indicate performance is higher than average. Higher scaled scores indicate better performance.
Time Frame: 13 weeks
Population: The analysis population comprises all individuals who signed an informed consent document and took at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | 9.13 (2.53) | 9.00 (1.87)

2. Primary Outcome: Controlled Oral Word Association Test
Description: The Controlled Oral Word Association Test is a measure of verbal fluency. Scores are standardized as z-scores (μ = 0, SD = 1) using age adjusted normative data provided by Tombaugh and Kozak (1996). A z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative z-scores indicate performance is lower than average, and positive z-scores indicate performance is higher than average. Positive z-scores indicate better performance.
Time Frame: 13 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | -0.35 (1.10) | -0.37 (0.93)

3. Primary Outcome: Stroop Interference Test
Description: The Stroop Interference Test is a measure of executive functioning. Scores are standardized as z-scores (μ = 0, SD = 1) using age adjusted normative data provided by PAR Incorporated (https://www.parinc.com/). A z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative z-scores indicate performance is lower than average, and positive z-scores indicate performance is higher than average. Positive z-scores indicate better performance.
Time Frame: 13 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | -0.15 (0.88) | -0.30 (0.96)

4. Primary Outcome: Symbol-Digit Modality Test
Description: The Symbol-Digit Modality Test is a measure of executive functioning. Scores are standardized as z-scores (μ = 0, SD = 1) using age adjusted normative data provided by WPS Publishers (https://www.wpspublish.com/). A z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative z-scores indicate performance is lower than average, and positive z-scores indicate performance is higher than average. Positive z-scores indicate better performance.
Time Frame: 13 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | 0.12 (0.82) | 0.05 (1.20)

5. Primary Outcome: Trail Making Test Part B
Description: The Trail Making Test Part B is a measure of executive functioning. Scores are standardized as z-scores (μ = 0, SD = 1) using age adjusted normative data provided by WPS Publishers (https://www.wpspublish.com/). A z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative z-scores indicate performance is lower than average, and positive z-scores indicate performance is higher than average. Positive z-scores indicate better performance.
Time Frame: 13 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | 0.01 (0.85) | -0.10 (1.35)

6. Secondary Outcome: Hopkins Verbal Learning Total Recall Test
Description: The Hopkins Verbal Learning Total Recall Test is an assessment of memory. Scores are standardized as T-scores (μ = 50, SD = 10) using age adjusted normative data provided by PAR Incorporated (https://www.parinc.com/). A T-score indicates the number of standard deviations away from the mean. A T-score of 50 is equal to the mean. T-scores below 50 indicate performance is lower than average, and T-scores above 50 indicate performance is higher than average. Higher T-scores indicate better performance.
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | 38.07 (8.92) | 39.57 (11.50)

7. Secondary Outcome: Semantic Fluency Test
Description: The Semantic Fluency Test is a measure of verbal fluency. Scores are standardized as z-scores (μ = 0, SD = 1) using age adjusted normative data provided by Tombaugh and Kozak (1996). A z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative z-scores indicate performance is lower than average, and positive z-scores indicate performance is higher than average. Positive z-scores indicate better performance.
Time Frame: 13 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 15 | 15
units on a scale | 0.41 (1.46) | -0.36 (0.95)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 20 weeks
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 12/15 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=15) | High Dose (N=15)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Low Dose (N=15) | High Dose (N=15)
Cold virus (Infections and infestations) | 1 (1) | 4 (4)
Short menstrual period (Reproductive system and breast disorders) | 1/14 (1) | 0/11 (0)
Menstrual cramps (Reproductive system and breast disorders) | 0/14 (0) | 1/11 (2)
Arm pain (General disorders) | 1 (1) | 0 (0)
Toothache (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataracts (Eye disorders) | 1 (1) | 0 (0)
Hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1)
Hemorrhoids (Renal and urinary disorders) | 1 (1) | 0 (0)
Poor appetite (General disorders) | 0 (0) | 1 (1)
Dark stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Strep throat (Infections and infestations) | 1 (1) | 0 (0)
Sore throat (General disorders) | 1 (3) | 0 (0)
Fall (Nervous system disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (1) | 0 (0)
Muscle aches (General disorders) | 0 (0) | 1 (1)
Goiter (Endocrine disorders) | 0 (0) | 1 (1)
Arhritis (General disorders) | 1 (1) | 1 (1)
Foot pain (General disorders) | 2 (2) | 0 (0)
Restlessness (General disorders) | 0 (0) | 1 (1)
Shoulder pain (General disorders) | 1 (1) | 0 (0)
Knee cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leg cramps (General disorders) | 2 (2) | 0 (0)
Motor vehicle accident (Social circumstances) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial experienced early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT02416193/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02416193/ICF_001.pdf